CLINICAL TRIAL: NCT05408676
Title: Comparison of Dexamethasone Alone vs in Combination With Pericardium 6 (P6) Electrical Stimulation or Granisetron in the Prevention of Postoperative Nausea and Vomiting in Patients Undergoing Breast Cancer Surgery
Acronym: P6 and PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jun Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2110244-11
Record Dates: First submitted 2022-05-30; First posted 2022-06-07 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Mammary Cancer; PONV
Keywords: Mammary Cancer; PONV; electric stimulation therapy; antiemetics
MeSH Terms: conditions — Breast Neoplasms; Postoperative Nausea and Vomiting | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Acu (Experimental): a surface electrode was applied in the induction room to the P6 acupoint on the dominant upper extremity, located ∼4 cm proximal to the distal wrist crease between the tendons of the flexor carpi radialis and the palmaris longus, and a negative surface electrode on the opposing dorsal aspect of the forearm. When the patient enters the operating room， an investigator connected the device to both electrodes with electrical wires, set initial electric stimulating current at 1 mA with the frequency at 2 Hz(square-wave pulses of 0.2 ms), gradually increased the current intensity until the patient felt pain or reached the discomfort threshold (ranging from 6 to 20 mA), and maintained the stimulation until end of operation.
  At the start of skin closure, saline (3 ml) was administered i.v.
  Interventions: Device: electric stimulation therapy
- Group Gra (Sham Comparator): Group Gra receive the same protocol but silicone covers were attached to both electrodesin to achieve an inert control.
  At the start of skin closure, granisetron (3 mg; Group Trp) was administered i.v.
  Interventions: Device: electric stimulation therapy
- Group Dxm (Sham Comparator): Group Dxm receive the same protocol but silicone covers were attached to both electrodesin to achieve an inert control.
  At the start of skin closure, saline (3 ml) was administered i.v.
  Interventions: Device: electric stimulation therapy

INTERVENTIONS:
Device: electric stimulation therapy — Transcutaneous electrical acupoint stimulation (TEAS) was achieved by an electrical neuromuscular stimulation device (JNR2; designed by the Department of Hand Surgery, Huashan Hospital, Fudan University, manufactured by Energy Conservation and Environment Protection Technology Company, Jiatong University, Shanghai,China)

SUMMARY:
Breast cancer is one of the three most common cancers worldwide, and the primary treatment method is surgery.Since most patients are non-smokers who use opioids in the postoperative period, which are known risk factors for postoperative nausea and vomiting (PONV) according to the Apfel Risk Score. Breast surgery was identified as a strong risk factor for PONV. According to the previous studies, the incidence of PONV is 30-70% in patients undergoing the breast cancer surgery, which not only gives patients unpleasant and painful experience, but also prolongs the hospital stays and delay patient discharge and adds to hospital costs. We compared the effects of dexamethasone alone vs. in combination with Pericardium 6 (P6) electrical stimulation or granisetron for inhibition of PONV in women undergoing breast cancer surgery.

DETAILED DESCRIPTION:
186 patients who are planed to undergo elective breast cancer surgery under general anaesthesia into the following three groups: acupoint stimulation+dexamethasone (Group Acu, n=62), granisetron +dexamethasone (Group Gra, n=62), and dexamethasone alone (Group Dxm, n=62). The incidence of nausea, vomiting, and need for rescue antiemetics was recorded 2, 6, 24, and 48 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing breast cancer resection under general anesthesia
* aged between 18 to 65
* American Society of Anesthesiologists grade I-II

Exclusion Criteria:

* using antiemetic drugs within 24 h before operation,
* nausea or vomiting within 24 h before operation;
* Alcoholic or drug abuse,
* abnormal liver and/or kidney function, diabetic or peripheral neuropathy patients, cardiovascular disease (excluding those with controlled hypertension).
* refuse to participate clinical trial

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
PONV within the first 24h after surgery | 24 hours after surgery.
  the incidence and severity of PONV

SECONDARY OUTCOMES:
PONV within the first 48h after surgery | 48 hours after surgery
  the incidence and severity of PONV
the use of postoperative antiemetics | 48 hours after surgery
  the frequency and dose of postoperative antiemetics
postoperative pain score | 3 months after surgery
  Numeric rating scale (NRS) at 2,6,24,48 hour and 3 month after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No